CLINICAL TRIAL: NCT04416399
Title: Use of High Dose Inhaled Corticosteroids as Treatment of Early COVID-19 Infection to Prevent Clinical Deterioration and Hospitalisation
Brief Title: STerOids in COVID-19 Study
Acronym: STOIC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Independent statistical review advice
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STOIC study
Record Dates: First submitted 2020-06-03; First posted 2020-06-04 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2020-07

CONDITIONS: Coronavirus Infection
Keywords: CoVID-19; Coronavirus infection; SARS-CoV-2
MeSH Terms: conditions — Coronavirus Infections; COVID-19 | interventions — Budesonide

STUDY DESIGN:
Intervention Model Description: Randomised, open label parallel group controlled clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Inhaled budesonide (Experimental): Budesonide inhaled via dry powder inhaler, 400 micrograms per inhalation, 2 inhalations twice a day
  Interventions: Drug: Budesonide dry powder inhaler
- Standard of care (No Intervention): Standard of care

INTERVENTIONS:
Drug: Budesonide dry powder inhaler — Budesonide inhaled via dry powder inhaler, 400 micrograms per inhalation, 2 inhalations twice a day
  Other Names: Pulmicort
  Arms: Inhaled budesonide

SUMMARY:
At the time of writing (3/4/2020), close to a million people have been infected by the SARS-CoV-2 coronavirus around the world. The severe clinical condition that leads to deaths is now called CoVID-19. Currently, there are no effective treatments for the early or late stages of this illness. Governments worldwide have undertaken dramatic interventions to try and reduce the rate of spread of this deadly coronavirus.

Early data from multiple studies in China, where the virus originated, show that severe cases of CoVID-19 are not as prevalent in patients with chronic lung diseases as expected. This data has been confirmed by the Italian physicians. The investigators think that the widespread use of inhaled corticosteroids reduces the risk of CoVID-19 pneumonia in patients with chronic lung disease. Early microbiological data also shows that these corticosteroids are effective at slowing down the rate of coronavirus replication on lung cells.

Inhaled corticosteroids are widely used to manage common lung conditions, such as asthma. This type of medicine is among the top 3 most common medication prescribed around the world. Their safety is well understood, and their potential side effects are mild and reversible.

The investigators propose to test this idea that, in participants early in the course of CoVID-19 illness, daily high dose inhaled corticosteroids for 28 days, will reduce the chances of severe respiratory illness needing hospitalisation. We will also study the effect of this inhaled therapy on symptoms and viral load.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the trial
* Male or Female, aged 18 years or above
* New onset of symptoms suggestive of COVID-19 e.g. new onset cough and/or fever, and/or loss of smell or taste within 7 or fewer days of participant being seen at visit 1
* In the Investigator's opinion, is able and willing to comply with all trial requirements

Exclusion Criteria:

* A known allergy to investigational medicine product (IMP) (budesonide)
* Any known contraindication to any of the IMPs (budesonide)
* Patient currently prescribed inhaled or systemic corticosteroids
* Recent use, within the previous 7 days of inhaled or systemic corticosteroids
* Patient needs hospitalisation at time of study consent
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.
* Participants who have participated in another research trial involving an investigational product in the past 12 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2020-07-16 (Actual); Primary Completion 2021-01-12 (Actual); Study Completion 2021-01-12 (Actual)

PRIMARY OUTCOMES:
Emergency department attendance of hospitalisation related to COVID-19 | Day 1 to day 28
  Evaluate the effect of intervention on emergency department attendance or hospitalisation related to COVID-19

SECONDARY OUTCOMES:
Body temperature | Day 1 to day 14
  Evaluate the effect of intervention on body temperature
Blood oxygen saturation level | Day 1 to day 14
  Evaluate the effect of intervention on blood oxygen level
Symptoms as assessed by common cold questionnaire | Day 1 to day 14
  Evaluate the effect of intervention on patient's symptoms as determined by common cold questionnaire. Higher score meaning worse symptoms.
Symptoms as assessed by FluPro questionnaire | Day 1 to day 14
  Evaluate the effect of intervention on patient's symptoms as determined by FluPro questionnaire. Higher score meaning worse symptoms.
Nasal/throat swab SARS-CoV-2 viral load | Day 1, 7 and 14
  Evaluate the effect of intervention on nasal and throat swab SARS-CoV-2 viral load

CONTACTS AND LOCATIONS:
Overall Officials: Mona Bafadhel, MBBS, PhD, Principal Investigator — University of Oxford
Locations (1):
- Oxford Respiratory Trials Unit, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cass SP, Nicolau DV Jr, Baker JR, Mwasuku C, Ramakrishnan S, Mahdi M, Barnes PJ, Donnelly LE, Martinez-Nunez RT, Russell REK, Bafadhel M. Coordinated nasal mucosa-mediated immunity accelerates recovery from COVID-19. ERJ Open Res. 2024 May 13;10(3):00919-2023. doi: 10.1183/23120541.00919-2023. eCollection 2024 May. PMID 38746861
- [Derived] Baker JR, Mahdi M, Nicolau DV Jr, Ramakrishnan S, Barnes PJ, Simpson JL, Cass SP, Russell REK, Donnelly LE, Bafadhel M. Early Th2 inflammation in the upper respiratory mucosa as a predictor of severe COVID-19 and modulation by early treatment with inhaled corticosteroids: a mechanistic analysis. Lancet Respir Med. 2022 Jun;10(6):545-556. doi: 10.1016/S2213-2600(22)00002-9. Epub 2022 Apr 7. PMID 35397798
- [Derived] Ramakrishnan S, Nicolau DV Jr, Langford B, Mahdi M, Jeffers H, Mwasuku C, Krassowska K, Fox R, Binnian I, Glover V, Bright S, Butler C, Cane JL, Halner A, Matthews PC, Donnelly LE, Simpson JL, Baker JR, Fadai NT, Peterson S, Bengtsson T, Barnes PJ, Russell REK, Bafadhel M. Inhaled budesonide in the treatment of early COVID-19 (STOIC): a phase 2, open-label, randomised controlled trial. Lancet Respir Med. 2021 Jul;9(7):763-772. doi: 10.1016/S2213-2600(21)00160-0. Epub 2021 Apr 9. PMID 33844996
- [Derived] Farne H, Singanayagam A. Reply. J Allergy Clin Immunol. 2021 Mar;147(3):1117-1118. doi: 10.1016/j.jaci.2020.11.019. Epub 2020 Dec 30. No abstract available. PMID 33388170
- [Derived] Nicolau DV, Bafadhel M. Inhaled corticosteroids in virus pandemics: a treatment for COVID-19? Lancet Respir Med. 2020 Sep;8(9):846-847. doi: 10.1016/S2213-2600(20)30314-3. Epub 2020 Jul 30. No abstract available. PMID 32738928